CLINICAL TRIAL: NCT02482792
Title: Norwegian Psychomotor Physiotherapy Versus Cognitive Patient Education and Active Physiotherapy
Brief Title: Norwegian Psychomotor Physiotherapy in Patients With Long-lasting Musculoskeletal Pain.
Acronym: NPMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tove Dragesund (Other)
Collaborators: Norwegian Fund for Postgraduate Training in Physiotherapy (Other)
Responsible Party: Sponsor-Investigator, Tove Dragesund, Post doc, University of Bergen
Organization: University of Bergen (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: d7k8fj2m
Record Dates: First submitted 2015-06-09; First posted 2015-06-26 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Physical Disability
Keywords: Musculoskeletal disorders; Psychosomatic; Pain
MeSH Terms: conditions — Musculoskeletal Diseases; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Norwegian Psychomotor Physiotherapy (Experimental): NPMP is a body-mind awareness approach, often given in a combination of massage, exercises and conversations. The NPMP is individualized, with duration of 45-60 minutes in each session. As the NPMP is a longitudinal and normally slow process to obtain change, treatment can last up till one year, in the beginning once a week, and after some time once a month.
  Interventions: Other: Norwegian Psychomotor Physiotherapy
- Cognitive Patient Education and PT (Active Comparator): The comparison group will receive a combination of education about how to manage pain (COPE) followed by active individual physiotherapy.They will receive one session weekly with COPE, given by a physiotherapist, maximum 4 times, followed by active individual Physiotherapy (PT).
  Interventions: Other: Cognitive Patient Education and PT

INTERVENTIONS:
Other: Norwegian Psychomotor Physiotherapy — The recruited patients will after randomization receive either Norwegian Psychomotor Physiotherapy (NPMP) or COPE combined with active individual physiotherapy. In NPMP the treatment is individualized, targeting body-mind awareness through exercise, massage and therapeutic conversation
  Other Names: NPMP
  Arms: Norwegian Psychomotor Physiotherapy
Other: Cognitive Patient Education and PT — The comparison group will receive a combination of education about how to manage pain (COPE) followed by active individual physiotherapy.
  Other Names: COPE- PT
  Arms: Cognitive Patient Education and PT

SUMMARY:
The aim is to examine the effect of Norwegian Psychomotor Physiotherapy (NPMP) in employees with long-lasting musculoskeletal pain compared to employees receiving Cognitive Patient Education in combination with active individual physiotherapy (COPE-PT) on pain, function, quality of life and sick-leave

DETAILED DESCRIPTION:
The NPMP is based on the assumption that patients with long-lasting problems, physical and/or psychological, may react with general aberrations related to posture, respiration, and movements, as well as with muscular tension and skin changes.

Employees With Long lasting musculoskeletal pain problems, working in the Municipality of Bergen, will be invited to participate in an Randomized Clinical Trial (RCT), and randomized to either receive Norwegian Psychomotor Physiotherapy (NPMP) or a series of Cognitive Patient Education in combination with active individual physiotherapy (COPE-PT). The aim is to examine the effect of NPMP compared to those receiving COPE-PT on pain, function, quality of life and sick-leave.

ELIGIBILITY:
Inclusion Criteria:

* Patients With neck,shoulder and/or widespread pain
* Pain (≥ 3 Numeric Pain Rating Scale (NPRS)
* Functional problems measured with Orebro Musculoskeletal Pain Screening Questionnaire (OMPSQ), Neck Disability Index (NDI) and/or Shoulder Pain and Disability Inventory (SPADI)-been sick-listed for 4-8 weeks, or on the brink of becoming sick-listed, or having had residual neck- and shoulder complaints problems during the last two years with several short-term sick-leaves.
* =/6 American College of Rheumatology (ACR) tender points,
* Reduced Relaxation and Flexibility from the Global Physiotherapy Examination (GPE)

Exclusion Criteria:

* Sick-listed > 6 months

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2017-10-26 (Actual)

PRIMARY OUTCOMES:
Efficacy of Norwegian Psychomotor Physiotherapy in Patients With Long-lasting pain | Change from baseline in pain at 3 months, at 6 months and 12 months.
  Pain on the Numeric Pain Rating Scale (NPRS)

SECONDARY OUTCOMES:
Efficacy of Norwegian Psychomotor Physiotherapy in Patients With Long-lasting pain | Change from baseline in wellbeing at 3 months, at 6 months and 12 months.
  Wellbeing on the Short Form-12 Health Survey (SF-12)
Efficacy of Norwegian Psychomotor Physiotherapy in Patients With Long-lasting pain | Change from baseline in sick-leave at 3 months, at 6 months and 12 months.
  Sick-leave
Efficacy of Norwegian Psychomotor Physiotherapy in Patients With Long-lasting pain | Change from baseline in shoulder function at 3 months, at 6 months and 12 months.
  Function on the Shoulder Pain and Disability Inventory (SPADI)
Efficacy of Norwegian Psychomotor Physiotherapy in Patients With Long-lasting pain | Change from baseline work related function at 3 months, at 6 months and 12 months.
  Function on the Norwegian Functional Assessment Scale (NFAS)
Efficacy of Norwegian Psychomotor Physiotherapy in Patients With Long-lasting pain | Change from baseline neck function at 3 months, at 6 months and 12 months.
  Neck Disability Index (NDI)
Efficacy of Norwegian Psychomotor Physiotherapy in Patients With Long-lasting pain | Change from baseline flexibility at 6 months.
  Global Body Examination-Flexibility (GBE)

CONTACTS AND LOCATIONS:
Overall Officials: Alice Kvåle, PhD, Principal Investigator — University of Bergen
Locations (1):
- Department of Global Public Health and Primary Care, UiB, Bergen, Hordaland, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dragesund T, Kvale A. Study protocol for Norwegian Psychomotor Physiotherapy versus Cognitive Patient Education in combination with active individualized physiotherapy in patients with long-lasting musculoskeletal pain - a randomized controlled trial. BMC Musculoskelet Disord. 2016 Aug 5;17:325. doi: 10.1186/s12891-016-1159-8. PMID 27496046